CLINICAL TRIAL: NCT00000572
Title: Extracorporeal Carbon Dioxide Removal for Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alan H. Morris, Professor, Director of Research, Pulmonary Division, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210; R01HL036787 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Acute Respiratory Distress Syndrome; Lung Diseases
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases | interventions — Positive-Pressure Respiration; Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extracorporeal membrane oxygenation (CO2 removal) (Experimental): Detailed Electronic Protocol Controlled Extracorporeal CO2 Removal with reduced positive-pressure ventilation
  Interventions: Procedure: extracorporeal membrane oxygenation (CO2 removal)
- Protocol Controlled positive-pressure vent (Active Comparator): Detailed Electronic Protocol Controlled positive-pressure ventilation
  Interventions: Procedure: positive-pressure ventilation

INTERVENTIONS:
Procedure: positive-pressure ventilation — Detailed computer protocol controlled positive pressure ventilation
  Arms: Protocol Controlled positive-pressure vent
Procedure: extracorporeal membrane oxygenation (CO2 removal) — Detailed computer protocol controlled Extracorporeal CO2 Removal with reduced positive pressure ventilation
  Arms: Extracorporeal membrane oxygenation (CO2 removal)

SUMMARY:
To compare conventional therapy using low frequency positive pressure ventilation with extracorporeal CO2 removal for the treatment of adult respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
BACKGROUND:

It is estimated that at least 150,000 individuals die each year of adult respiratory distress syndrome. Treatment remains largely supportive. The National Heart, Lung, and Blood Institute (NHLBI) conducted the Extracorporeal Support for Respiratory Insufficiency (ECMO, Extracorporeal Membrane Oxygenation) trial from June 1974 through 1978. In ECMO, 90 patients were randomized to either extracorporeal membrane oxygenation plus conventional therapy or to conventional therapy. Survival rates were less than ten percent in both groups. The failure of the trial to demonstrate the superiority of ECMO over conventional ventilatory support resulted in the virtual elimination of the use of ECMO in clinical medicine.

In the earlier NHLBI trial, ECMO was implemented with a veno-arterial shunt which approximated 90 percent of the baseline cardiac output. Ventilation of the lungs was continued with reduced function of inspiration oxygen. Thus, the lungs were deprived of the principle source of blood supply while continuously exposed to potentially injurious ventilatory pressures and gas composition. The present patient trial used a new form of therapy developed by Dr. Gattinoni and co-workers in Milan, Italy with the collaboration of Dr. Kolobow at the National Institutes of Health in Bethesda. The authors reported a 77 percent survival rate for the new therapy. In Step 1 of the new therapy, the patient was initially ventilated with pressure-controlled, inverted ratio ventilation. If the patient did not improve, Step 2 using extracorporeal perfusion was performed with a veno-venous shunt in contrast to a veno-arterial shunt. The veno-venous shunt preserved pulmonary blood flow whereas the veno-arterial shunt diminished it. Step 3 was reserved for those patients who did not meet the therapeutic criteria of Step 2. They underwent low frequency positive-pressure ventilation and extracorporeal CO2 removal involving veno-venous bypass via the internal jugular and femoral or bilateral saphenous veins.

DESIGN NARRATIVE:

Randomized, fixed sample. Patients were stratified by age (under and over 40 years) and by the presence or absence of trauma. Patients were assigned to conventional positive pressure ventilation therapy or to a three-step therapeutic program employing pressure-controlled-inverted-ratio-ventilation, continuous positive airway pressure, and low-frequency positive pressure ventilation-extracorporeal CO2 removal. The main outcome measure was survival at 30 days after randomization. Secondary outcome measures included hospital costs, physiologic data, length of hospital stay, and blood product consumption. Follow-up took place during the year after hospital discharge.

ELIGIBILITY:
Men and women with acute respiratory distress syndrome.

Inclusion Criteria: ECMO ENTRY CRITERIA (PaO2 < 50 mm Hg -REPEATED THREE TIMES):

Rapid entry: 2 hours at fraFIO2=1.00 and PEEP>5 cm H2O with PaCO2=30-45 mmHg

Slow entry: 12 hours at fraction of inspired oxygen (FIO2)>0.60 and positive end-expiratory pressure (PEEP)>5 cm H2O with PaCO2=30-45 mmHg and right to Left shunt fraction >0.30

Exclusion Criteria:

1. Contraindication to anti-coagulation (for example, gastrointestinal bleeding, recent cerebrovascular accident, or chronic bleeding disorder).
2. Pw > 25 mm Hg (superseded by our screening criterion that Pw ~ 15 mm Hg).
3. Mechanical ventilation >21. days.
4. Severe chronic systemic disease or another clinical condition that, in itself,greatly limits survival; for example,

   1. Irreversible central nervous system disease
   2. Severe chronic pulmonary disease (forced expiratory volume in 1 second (FEV1)<1 L, FEV1/FVC(forced vital capacity) <0.3 of predicted, chronic PaCO2 >45 mm Hg, chest x-ray evidence of overinflation or interstitial infiltration, or previous hospitalization for chronic respiratory insufficiency)
   3. Total-body surface burns> 40%
   4. Rapidly fatal malignancy
   5. Chronic left ventricular failure
   6. Chronic renal failure (we required serum creatlnlne ~ 2 mg/dl or chronic dialysis therapy)
   7. Chronic liver failure (we required total serum bilirubin;?; 2 mg/dl)
   8. Immunosuppressed patients and patients with a positive human immu.. nodeficiency virus test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1987-06; Primary Completion 1991-04 (Actual); Study Completion 1993-01 (Actual)

PRIMARY OUTCOMES:
Survival | Hospital stay (time until death): participants will be followed for the duration of hospital stay, an expected average of 30 days).
  All deaths occurred within 30 days of enrollment

SECONDARY OUTCOMES:
Hospital days | up to hospital discharge, approximately 30 days
ICU days | up to ICU discharge, approximately 30 days

OTHER OUTCOMES:
Hospital costs | Hospital stay
  $US
Bleeding/Hemorrhage | Hospital stay
  Bleeding in ECCO2R subjects exceeded that in control subjects

REFERENCES:
- [Background] Morris AH, Menlove RL, Rollins RJ, Wallace CJ, Beck E. A controlled clinical trial of a new 3-step therapy that includes extracorporeal CO2 removal for ARDS. ASAIO Trans. 1988 Jan-Mar;34(1):48-53. No abstract available. PMID 3132189
- [Background] Sittig DF, Gardner RM, Pace NL, Morris AH, Beck E. Computerized management of patient care in a complex, controlled clinical trial in the intensive care unit. Comput Methods Programs Biomed. 1989 Oct-Nov;30(2-3):77-84. doi: 10.1016/0169-2607(89)90060-6. PMID 2684495
- [Background] Sittig DF, Pace NL, Gardner RM, Beck E, Morris AH. Implementation of a computerized patient advice system using the HELP clinical information system. Comput Biomed Res. 1989 Oct;22(5):474-87. doi: 10.1016/0010-4809(89)90040-2. PMID 2776450
- [Background] Sittig DF, Gardner RM, Morris AH, Wallace CJ. Clinical evaluation of computer-based respiratory care algorithms. Int J Clin Monit Comput. 1990 Jul;7(3):177-85. doi: 10.1007/BF02915583. PMID 2250128
- [Background] Suchyta MR, Elliott CG, Colby T, Rasmusson BY, Morris AH, Jensen RL. Open lung biopsy does not correlate with pulmonary function after the adult respiratory distress syndrome. Chest. 1991 May;99(5):1232-7. doi: 10.1378/chest.99.5.1232. PMID 2019184
- [Background] Suchyta MR, Clemmer TP, Orme JF Jr, Morris AH, Elliott CG. Increased survival of ARDS patients with severe hypoxemia (ECMO criteria). Chest. 1991 Apr;99(4):951-5. doi: 10.1378/chest.99.4.951. PMID 2009801
- [Background] Henderson S, Crapo RO, Wallace CJ, East TD, Morris AH, Gardner RM. Performance of computerized protocols for the management of arterial oxygenation in an intensive care unit. Int J Clin Monit Comput. 1991-1992;8(4):271-80. doi: 10.1007/BF01739128. PMID 1820417
- [Background] East TD, Morris AH, Wallace CJ, Clemmer TP, Orme JF Jr, Weaver LK, Henderson S, Sittig DF. A strategy for development of computerized critical care decision support systems. Int J Clin Monit Comput. 1991-1992;8(4):263-9. doi: 10.1007/BF01739127. PMID 1820416
- [Background] Suchyta MR, Clemmer TP, Elliott CG, Orme JF Jr, Weaver LK. The adult respiratory distress syndrome. A report of survival and modifying factors. Chest. 1992 Apr;101(4):1074-9. doi: 10.1378/chest.101.4.1074. PMID 1555423
- [Background] East TD, Bohm SH, Wallace CJ, Clemmer TP, Weaver LK, Orme JF Jr, Morris AH. A successful computerized protocol for clinical management of pressure control inverse ratio ventilation in ARDS patients. Chest. 1992 Mar;101(3):697-710. doi: 10.1378/chest.101.3.697. PMID 1541135
- [Background] Morris AH, East TD, Wallace CJ, Orme J Jr, Clemmer T, Weaver L, Thomas F, Dean N, Pearl J, Rasmusson B. Ethical implications of standardization of ICU care with computerized protocols. Proc Annu Symp Comput Appl Med Care. 1994:501-5. PMID 7949979
- [Background] Morris AH. Adult respiratory distress syndrome and new modes of mechanical ventilation: reducing the complications of high volume and high pressure. New Horiz. 1994 Feb;2(1):19-33. PMID 7922426
- [Background] Morris AH. Uncertainty in the management of ARDS: lessons for the evaluation of a new therapy. Intensive Care Med. 1994;20(2):87-9. doi: 10.1007/BF01707658. No abstract available. PMID 8201102
- [Background] Suchyta MR, Elliott CG, Jensen RL, Crapo RO. Predicting the presence of pulmonary function impairment in adult respiratory distress syndrome survivors. Respiration. 1993;60(2):103-8. doi: 10.1159/000196182. PMID 8341851
- [Background] Morris AH. Protocol management of adult respiratory distress syndrome. New Horiz. 1993 Nov;1(4):593-602. PMID 8087579
- [Result] Morris AH, Wallace CJ, Menlove RL, Clemmer TP, Orme JF Jr, Weaver LK, Dean NC, Thomas F, East TD, Pace NL, Suchyta MR, Beck E, Bombino M, Sittig DF, Bohm S, Hoffmann B, Becks H, Butler S, Pearl J, Rasmusson B. Randomized clinical trial of pressure-controlled inverse ratio ventilation and extracorporeal CO2 removal for adult respiratory distress syndrome. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):295-305. doi: 10.1164/ajrccm.149.2.8306022.
- [Result] Habashi NM, Reynolds HN, Borg U, Cowley RA. Randomized clinical trial of pressure-controlled inverse ration ventilation and extra corporeal CO2 removal for ARDS. Am J Respir Crit Care Med. 1995 Jan;151(1):255-6. doi: 10.1164/ajrccm.151.1.7812567. No abstract available.
- [Result] Brunet F, Mira JP, Dhainaut JF, Dall'ava-Santucci J. Efficacy of low-frequency positive-pressure ventilation-extracorporeal CO2 removal. Am J Respir Crit Care Med. 1995 Apr;151(4):1269-70. doi: 10.1164/ajrccm/151.4.1269-a. No abstract available. PMID 7697266
- [Result] Falke KJ. Randomized clinical trial of pressure-controlled inverse ratio ventilation and extracorporeal CO2 removal for adult respiratory distress syndrome. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):1016-7. No abstract available. PMID 9310029